CLINICAL TRIAL: NCT01595152
Title: Solifenacin Succinate vs. Fesoterodine A Comparison Trial for the Treatment of Bothersome Urgency Symptoms
Brief Title: Solifenacin Succinate Versus Fesoterodine A Comparison Trial for Urgency Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Lior Lowenstein, Head Of Urgoyncology Service, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMB-0096-12; RMB-0096-12 (Other: Helsinki Rambam)
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Urinary Bladder, Overactive
Keywords: Urgency, urgency incontinence,USIQ
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; fesoterodine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- solifenacin succinate (10 mg OD) (Active Comparator)
  Interventions: Drug: solifenacin succinate
- fesoterodine (8mg OD) (Active Comparator)
  Interventions: Drug: fesoterodine

INTERVENTIONS:
Drug: solifenacin succinate — 8 mg once daily for 60 days
  Other Names: vesicare
  Arms: solifenacin succinate (10 mg OD)
Drug: fesoterodine — 8 mg, once daily for 60 dyas
  Other Names: Toviaz
  Arms: fesoterodine (8mg OD)

SUMMARY:
Hypothesis:

Objective 1: To advance the investigators understanding on the effect of solifenacin succinate (10 mg OD) vs. fesoterodine (8mg OD) on urinary urgency using a validated Urgency Severity and Impact Questionnaire (USIQ).

Hypothesis 1.1: The severity of urgency symptoms as measured by USIQ will change differently in women with OAB following a 3 month treatment with solifenacin succinate (10 mg OD) vs. fesoterodine (8mg OD).

Hypothesis 2.1: Condition-specific quality of life (QOL) as measured by USIQ will change differently in women with OAB following a 3 month treatment with solifenacin succinate (10 mg OD) vs. fesoterodine (8mg OD).

Objective 2: To advance the investigators understanding on the adverse events (AE's) of solifenacin succinate (10 mg OD) vs. fesoterodine (8mg OD).

Hypothesis 1.1: The severity and rate of AE's in women with OAB following a 3 month of treatment with solifenacin succinate (10 mg OD) vs. fesoterodine (8mg OD) will be different.

DETAILED DESCRIPTION:
The National Overactive Bladder Evaluation (NOBLE) Program estimated the prevalence of OAB in the US is nearly 17% affecting approximately 30 million adults. Sixty-one percent of adults with OAB also have urge urinary incontinence (UUI. Urinary urgency is a key symptom of OAB. Urgency may be more bothersome to patients than urinary frequency, although urinary frequency is often the primary focus of study in the field of OAB. This may be partially due to controversy surrounding how to define the term 'urinary urgency'. As currently defined, urgency is meant to describe an abnormal sensation that is distinguishable from the normal feeling of "urge to void," which occurs during a normal bladder-filling cycle. Attempts to measure urgency are confounded by difficulties in understanding this definition in the context of a normal "urge" to void. This controversy probably arises because of the overlap of the English words 'urge' and 'urgency' during clinical conversation, and apparently does not give rise to confusion in other languages. Recently a new validated questionnaire for the measurement of urgency symptoms was validated[5, 6]. The USIQ consists of two parts with an initial filter question, designated for self-administration. The first 5 items, known as USIQ- severity (USIQ-S), inquires about urgency symptoms and severity, while the second part USIQ- quality of life (USIQ-QOL) consists of 8 questions which inquire about bother and condition specific QOL such as: cooping behaviors, work, commuting and travel, sleep, physical activities, social activities, psychological well-being, relationships and sexual function. Items for each scale are summed and transformed to a score ranging from 0-100. Higher symptom bother scores indicate increasing symptom bother, and higher USIQ-QOL scores indicate worse health related quality of life. The main objective of this current study is to compare the effect of two different anticholinergic medications on symptoms of urinary urgency using a validated, subjective instruments designed specifically for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* Are > 18 years old
* Have a clinical diagnosis of OAB (wet or dry) with urinary urgency
* Are seeking treatment for OAB
* No contraindication to solifenacin succinate (10 mg OD) or fesoterodine (8mg OD)
* Have a negative urine dipstick analysis
* Are able to consent and fill out study documents and complete all study visits
* Have not been treated with an anticholinergic medication in the past 1-month

Exclusion Criteria:

* Have known neurologic disorder, e.g.: multiple sclerosis, Parkinson's Disease, spinal cord injury, stroke
* Are currently receiving treatment for OAB, including medications, physical and/or formal behavioral therapy, or electrical stimulation
* Have an elevated post -void residual volume by ultrasound or straight catheterization (PVR>150 ml)
* Were treated for a urinary tract infection in the last month
* Have untreated narrow angle glaucoma
* Are unable to comprehend and complete study tasks
* Have an allergy to or had previously failed treatment with solifenacin succinate or fesoterodine

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Changes in urgency sensation | two months following treatment
  The effect of two different antochloinergic treatment on urgency symptoms will be measured by comparing USIQ scores changes in the two study arms, before and after treatment. Changes in urgency sensation will be analysed by subsiding the USIQ scopre at 2 months (second visit) from the USIQ score at baseline. Independent student t- test will be used for Comparison between the changes in USIQ score of the two groups.

SECONDARY OUTCOMES:
Adverse events | two months
  Tolerability of both drugs will be monitored throughout the study based on reported AEs and discontinuations.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Padoa, MD, Principal Investigator — Assaf-Harofeh Medical Center; Haim Krissi, MD, Principal Investigator — Belinson Medical center; David Shveiky, MD, Principal Investigator — Hadassa; Naama Marcus, MD, Principal Investigator — Rebecca ziv; Lior Lowenstein, MD, MS, Principal Investigator — Rambam Health Care Campus
Locations (5):
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah, Jerusalem
  - Belinson, Petah Tikva
  - Rebecca Ziv, Safed
  - Asaf harofeh, Tel Aviv